CLINICAL TRIAL: NCT00714987
Title: Predictive Value of the Extra-Vascular Lung Water (EVLW) for the Alveolar Recruitment in the Acute Respiratory Distress Syndrome ( ARDS ).
Brief Title: The EVLW for Set the Positive End Expiratory Pressure (PEEP) in the Acute Respiratory Distress Syndrome (ARDS)
Status: Withdrawn | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, directeur Adjoint, Organization: University Hospital, Strasbourg, France
Other Study IDs: 3800
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Mechanical ventilation; PEEP with low level; PEEP with high level; EVLW; Picco® system; PaO2/FiO2 ratio
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: High level PEEP
- 2: Low level PEEP

SUMMARY:
* ARDS is a severe pathology with high mortality and morbidity.Actual ventilatory management is clear for the set of the tidal volume and for the survey of the plateau pressure for the patients who require mechanical ventilation.
* The set of the PEEP (low or high levels) remains unclear : it seems that some patients need low levels of PEEP whereas anther need high levels; but there is no validated data that can discriminate them.
* We hypothesized that patients with low levels of EVLW ( measured with the Picco® system ) need low level of PEEP to ameliorate their oxygenation ( measured with the PaO2/FiO2 ratio ) whereas patients with high levels of EVLW) need high levels of PEEP.

ELIGIBILITY:
Inclusion Criteria:

* age>18;
* ARDS criteria.

Exclusion Criteria:

* severe pulmonary hypertension;
* chronic right ventricular failure;
* pulmonary embolism;
* tricuspidian valvulopathy;
* history of spontaneous pneumothorax;
* severe emphysema;
* bronchomalacia;
* recent pulmonary surgery;
* BMI>40;
* Interstitial pulmonary fibrosis;
* End of life;
* Chronic neuromyopathie;
* Recent neurosurgery or intracranian hypertension;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients mechanically ventilated, monitored with the Picco® system, hospitalized in a medical critical care unit of an university hospital
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Estimate the Lung Water Extra-Vascular as predictive marker of the answer (Variation of needs in oxygen) to the ventilatory strategy: the low level, and high level of pressure positive expiratory, in the SDRA | During all the period of stay of the patient Intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Fady KARA, MD, Principal Investigator — University Hospital, Strasbourg, France